CLINICAL TRIAL: NCT04794413
Title: An Open Label, Proof-of-Principle, Pilot Study to Evaluate Pimavanserin for the Treatment of Motor and Behavioral Symptoms of Tourette Syndrome
Brief Title: Pimavanserin Treatment in TS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joseph Jankovic (Other)
Collaborators: Andrew Billnitzer, MD (Unknown)
Responsible Party: Sponsor-Investigator, Joseph Jankovic, Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43658
Record Dates: First submitted 2021-03-02; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Tourette Syndrome; Tardive Dyskinesia
Keywords: pimavanserin; Tourette Syndrome; tics
MeSH Terms: conditions — Tourette Syndrome; Tardive Dyskinesia; Tics | interventions — pimavanserin

STUDY DESIGN:
Intervention Model Description: This is an open-label, proof-of-principle, 8-week treatment, pilot study for male and female patients aged 18 years and older with Tourette Syndrome. There were no control groups nor randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pimavanserin (Experimental): All participants will receive pimavanserin 17mg once daily for 1 week and, if the tics are deemed to be inadequately controlled then increase to 34 mg once daily, taken orally as two 17 mg tablets once daily.
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin is a serotonin receptor inverse agonist used in treatment of psychosis in Parkinson's disease.
  Other Names: Nuplazid

SUMMARY:
This research study is determining if a drug called Pimavanserin if safe and effective in the treatment of the symptoms of Tourette Syndrome. Pimavanserin is an investigational drug for Tourette Syndrome, which means it has not been approved by the United States Food and Drug Administration (FDA) to treat Tourette Syndrome. Pimavanserin has been approved by the FDA as a treatment for hallucinations in Parkinson's Disease. It is currently marketed under the name NUPLAZID (pimavanserin) capsules by Acadia Pharmaceuticals.

DETAILED DESCRIPTION:
Tourette Syndrome is typically treated with drugs that block or reduce the function of dopamine (a brain chemical involved in movement). However, many of these drugs have adverse effects including irreversible, involuntary movements, typically affecting the face, known as tardive dyskinesia. Newer drugs may have lower risk of tardive dyskinesia. However, many of these drugs are still in clinical trials or are very expensive when used off-label (without FDA approval) to treat Tourette Syndrome. Given these limitations, exploring the potential of other drugs is essential in helping patients.

Several studies have shown that serotonin, another chemical in the brain like dopamine, may also play a role in the symptoms of Tourette Syndrome. Serotonin is already the target of many drugs in the treatment of depression, anxiety and obsessive-compulsive disorder which frequently occur in patients with Tourette Syndrome. Pimavanserin is also a drug that works on serotonin system. This means it may be helpful in the treatment of Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients meet the Diagnostic and Statistical Manuel of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for TS and, in the opinion of the investigator and patient, the patient's active tics are causing distress or impairment.
* Patient has a TTS of 20 or higher on the YGTSS at screening and baseline.
* Patient can swallow study medical whole.
* Patient is willing to adhere to the medication regimen and to comply with all study procedures.
* Patient is in good general health, as indicated by the medical and psychiatric history as well as physical and neurological examination.
* In the investigator's opinion, the patient has the ability to understand the nature of the study and its procedures, and the patient is expected to complete the study as designed.
* Patient has provided written informed consent according to local regulations.
* Females who are postmenarchal or greater than 12 years of age may be included if they have a negative urine pregnancy test at baseline or are sterile.
* Females who are postmenarchal or great than 12 years of age who male partners are potentially fertile (i.e. no vasectomy) must use highly effective birth control methods for the duration of the study (i.e. starting at screening) and for 30 days or 5 half-lives, whichever is longer after last dose of pimavanserin. The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

* Patient has a neurological disorder other than TS that could obscure the evaluation of tics.
* The patient's predominant movement disorder is stereotypy (coordinated movements that repeat continually and identically) associated with autism spectrum disorder.
* Patient has a confirmed diagnosis of bipolar disorder, schizophrenia, or another psychotic disorder.
* Patient has a DSM diagnosis at screening that, in the opinion of the investigator, makes the patient unsuitable for the study.
* Patient has received Comprehensive Behavioral Intervention for Tics for TS or Cognitive Behavioral Therapy for OCD within 4 weeks of screening.
* Patient has received treatment with deep brain stimulation, transmagnetic stimulation, or transcranial direct current stimulation within 4 weeks of the screening visit for reduction of tics.
* Stroke or other uncontrolled serious medical illness such as myocardial infarction within 6 months of baseline.
* Patient with unknown QT prolongation or in combination with other drugs known to prolong QT interval including Class 1A antiarrhythmics (e.g., quinidine, procainamide) or Class 3 antiarrhythmics (e.g., amiodarone, sotalol), certain antipsychotics medications (e.g., ziprasidone, chlorpromazine, thioridazine), and certain antibiotics (e.g., gatifloxacin, moxifloxacin).
* Patients with a history of cardiac arrhythmias, as well as other circumstances that may increase the risk of the occurrence of torsade de pointes and/or sudden death, including symptomatic bradycardia, hypokalemia or hypomagnesemia, and the presence of congenital prolongation of the QT interval.
* Patient has evidence of hepatic impairment.
* Patient has a known allergy to any of the components of pimavanserin.
* Patient has participated in an investigational drug or device study and received intervention within 30 days or 5 drug half-lives of baseline, whichever is longer.
* Patient is a pregnant or lactating female, or plans to be pregnant during the study.
* Patient has a history of or acknowledges alcohol-related disorder in the previous 12 months, as defined in the DSM-5.
* Patient has a positive urine drug screen test result or is unable to refrain from substance abuse throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of pimavanserin on Tourette Syndrome | 10 weeks
  The primary objective is to evaluate the effect of pimavanserin on motor and phonic tics associated with Tourette Syndrome using the Yale Global Tic Severity Scale. The minimum score for this scale is 0 and the maximum score for this scale 100. A higher score suggests a more sever Tic or that the Tic has a greater impact on the person's life.

SECONDARY OUTCOMES:
Evaluate the effect of pimavanserin on Tourette Syndrome | 10 weeks
  A secondary objective is to evaluate the effect of pimavanserin on obsessive-compulsive behaviors associated with Tourette Syndrome using the Yale-Brown Obsessive Compulsive Scale. The minimum score of this scale is 0 and the maximum score of this scale is 40. A higher score represents greater severity of obsessive compulsive symptoms.
Evaluate the effect of pimavanserin on Tourette Syndrome | 10 weeks
  A secondary objective is to evaluate the effect of pimavanserin on motor and phonic tics associated with Clinical Global Impression Scale. The minimum score of this scale is 1 and the maximum score of this scale is 7. A higher score suggests a more sever symptom.
Evaluate the effect of pimavanserin on Tourette Syndrome | 10 weeks
  A secondary objective is to evaluate the effect of pimavanserin on motor and phonic tics associated with Patient Global Impression of Improvement Scale. The minimum score of this scale is 1 and the maximum score of this scale is 7. A higher score suggests symptoms are very much worse.
Evaluate the effect of pimavanserin on Tourette Syndrome | 10 weeks
  A secondary objective is to evaluate the effect of pimavanserin on motor and phonic tics and obsessive-compulsive behaviors associated with Tourette Syndrome using the Columbia-Suicide Severity Rating Scale (C-SSRS). The minimum score of this scale is 2 and the maximum score of this scale is 25, with a higher score indicating more intense ideation and greater risk.
Evaluate the effect of pimavanserin on Tourette Syndrome | 10 weeks
  A secondary objective is to evaluate the effect of pimavanserin on motor and phonic tics and obsessive-compulsive behaviors associated with Tourette Syndrome using the Gilles de la Tourette Syndrome Quality of Life Scale. The minimum score is 0 and the maximum score is 108, with a higher score indicating extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.

REFERENCES:
- [Background] Jankovic J, Kurlan R. Tourette syndrome: evolving concepts. Mov Disord. 2011 May;26(6):1149-56. doi: 10.1002/mds.23618. Epub 2011 Apr 11. PMID 21484868
- [Background] Thenganatt MA, Jankovic J. Recent Advances in Understanding and Managing Tourette Syndrome. F1000Res. 2016 Feb 9;5:F1000 Faculty Rev-152. doi: 10.12688/f1000research.7424.1. eCollection 2016. PMID 26918185
- [Background] Billnitzer A, Jankovic J. Current Management of Tics and Tourette Syndrome: Behavioral, Pharmacologic, and Surgical Treatments. Neurotherapeutics. 2020 Oct;17(4):1681-1693. doi: 10.1007/s13311-020-00914-6. PMID 32856174
- [Background] Robertson MM, Eapen V, Singer HS, Martino D, Scharf JM, Paschou P, Roessner V, Woods DW, Hariz M, Mathews CA, Crncec R, Leckman JF. Gilles de la Tourette syndrome. Nat Rev Dis Primers. 2017 Feb 2;3:16097. doi: 10.1038/nrdp.2016.97. PMID 28150698
- [Background] Paschou P, Fernandez TV, Sharp F, Heiman GA, Hoekstra PJ. Genetic susceptibility and neurotransmitters in Tourette syndrome. Int Rev Neurobiol. 2013;112:155-77. doi: 10.1016/B978-0-12-411546-0.00006-8. PMID 24295621
- [Background] Udvardi PT, Nespoli E, Rizzo F, Hengerer B, Ludolph AG. Nondopaminergic neurotransmission in the pathophysiology of Tourette syndrome. Int Rev Neurobiol. 2013;112:95-130. doi: 10.1016/B978-0-12-411546-0.00004-4. PMID 24295619
- [Background] Forde NJ, Kanaan AS, Widomska J, Padmanabhuni SS, Nespoli E, Alexander J, Rodriguez Arranz JI, Fan S, Houssari R, Nawaz MS, Rizzo F, Pagliaroli L, Zilhao NR, Aranyi T, Barta C, Boeckers TM, Boomsma DI, Buisman WR, Buitelaar JK, Cath D, Dietrich A, Driessen N, Drineas P, Dunlap M, Gerasch S, Glennon J, Hengerer B, van den Heuvel OA, Jespersgaard C, Moller HE, Muller-Vahl KR, Openneer TJ, Poelmans G, Pouwels PJ, Scharf JM, Stefansson H, Tumer Z, Veltman DJ, van der Werf YD, Hoekstra PJ, Ludolph A, Paschou P. TS-EUROTRAIN: A European-Wide Investigation and Training Network on the Etiology and Pathophysiology of Gilles de la Tourette Syndrome. Front Neurosci. 2016 Aug 23;10:384. doi: 10.3389/fnins.2016.00384. eCollection 2016. PMID 27601976
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Cavanna AE, Schrag A, Morley D, Orth M, Robertson MM, Joyce E, Critchley HD, Selai C. The Gilles de la Tourette syndrome-quality of life scale (GTS-QOL): development and validation. Neurology. 2008 Oct 28;71(18):1410-6. doi: 10.1212/01.wnl.0000327890.02893.61. PMID 18955683
- [Background] Jeon S, Walkup JT, Woods DW, Peterson A, Piacentini J, Wilhelm S, Katsovich L, McGuire JF, Dziura J, Scahill L. Detecting a clinically meaningful change in tic severity in Tourette syndrome: a comparison of three methods. Contemp Clin Trials. 2013 Nov;36(2):414-20. doi: 10.1016/j.cct.2013.08.012. Epub 2013 Aug 31. PMID 24001701
- [Background] Rothenberger A, Roessner V. Psychopharmacotherapy of Obsessive-Compulsive Symptoms within the Framework of Tourette Syndrome. Curr Neuropharmacol. 2019;17(8):703-709. doi: 10.2174/1570159X16666180828095131. PMID 30152283
- [Background] McDougle CJ, Goodman WK, Leckman JF, Barr LC, Heninger GR, Price LH. The efficacy of fluvoxamine in obsessive-compulsive disorder: effects of comorbid chronic tic disorder. J Clin Psychopharmacol. 1993 Oct;13(5):354-8. PMID 8227493
- [Background] Leckman JF, Goodman WK, Anderson GM, Riddle MA, Chappell PB, McSwiggan-Hardin MT, McDougle CJ, Scahill LD, Ort SI, Pauls DL, et al. Cerebrospinal fluid biogenic amines in obsessive compulsive disorder, Tourette's syndrome, and healthy controls. Neuropsychopharmacology. 1995 Feb;12(1):73-86. doi: 10.1038/sj.npp.1380241. PMID 7766289
- [Background] Comings DE. Blood serotonin and tryptophan in Tourette syndrome. Am J Med Genet. 1990 Aug;36(4):418-30. doi: 10.1002/ajmg.1320360410. PMID 2389798
- [Background] Cath DC, Spinhoven P, Landman AD, van Kempen GM. Psychopathology and personality characteristics in relation to blood serotonin in Tourette's syndrome and obsessive-compulsive disorder. J Psychopharmacol. 2001 Jun;15(2):111-9. doi: 10.1177/026988110101500208. PMID 11448084
- [Background] Higgins GA, Enderlin M, Haman M, Fletcher PJ. The 5-HT2A receptor antagonist M100,907 attenuates motor and 'impulsive-type' behaviours produced by NMDA receptor antagonism. Psychopharmacology (Berl). 2003 Nov;170(3):309-319. doi: 10.1007/s00213-003-1549-0. Epub 2003 Aug 7. PMID 12904968
- [Background] Wong DF, Brasic JR, Singer HS, Schretlen DJ, Kuwabara H, Zhou Y, Nandi A, Maris MA, Alexander M, Ye W, Rousset O, Kumar A, Szabo Z, Gjedde A, Grace AA. Mechanisms of dopaminergic and serotonergic neurotransmission in Tourette syndrome: clues from an in vivo neurochemistry study with PET. Neuropsychopharmacology. 2008 May;33(6):1239-51. doi: 10.1038/sj.npp.1301528. Epub 2007 Nov 7. PMID 17987065
- [Background] Haugbol S, Pinborg LH, Regeur L, Hansen ES, Bolwig TG, Nielsen FA, Svarer C, Skovgaard LT, Knudsen GM. Cerebral 5-HT2A receptor binding is increased in patients with Tourette's syndrome. Int J Neuropsychopharmacol. 2007 Apr;10(2):245-52. doi: 10.1017/S1461145706006559. Epub 2006 Feb 28. PMID 16945163
- [Background] Steeves TD, Fox SH. Neurobiological basis of serotonin-dopamine antagonists in the treatment of Gilles de la Tourette syndrome. Prog Brain Res. 2008;172:495-513. doi: 10.1016/S0079-6123(08)00924-2. PMID 18772048
- [Background] McCracken JT, Suddath R, Chang S, Thakur S, Piacentini J. Effectiveness and tolerability of open label olanzapine in children and adolescents with Tourette syndrome. J Child Adolesc Psychopharmacol. 2008 Oct;18(5):501-8. doi: 10.1089/cap.2007.135. PMID 18928414
- [Background] Weisman H, Qureshi IA, Leckman JF, Scahill L, Bloch MH. Systematic review: pharmacological treatment of tic disorders--efficacy of antipsychotic and alpha-2 adrenergic agonist agents. Neurosci Biobehav Rev. 2013 Jul;37(6):1162-71. doi: 10.1016/j.neubiorev.2012.09.008. Epub 2012 Oct 23. PMID 23099282
- [Background] Porta M, Sassi M, Cavallazzi M, Fornari M, Brambilla A, Servello D. Tourette's syndrome and role of tetrabenazine: review and personal experience. Clin Drug Investig. 2008;28(7):443-59. doi: 10.2165/00044011-200828070-00006. PMID 18544005
- [Background] Jankovic J, Jimenez-Shahed J, Budman C, Coffey B, Murphy T, Shprecher D, Stamler D. Deutetrabenazine in Tics Associated with Tourette Syndrome. Tremor Other Hyperkinet Mov (N Y). 2016 Nov 7;6:422. doi: 10.7916/D8M32W3H. eCollection 2016. PMID 27917309
- [Background] Bonnier C, Nassogne MC, Evrard P. Ketanserin treatment of Tourette's syndrome in children. Am J Psychiatry. 1999 Jul;156(7):1122-3. doi: 10.1176/ajp.156.7.1122a. No abstract available. PMID 10401479

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04794413/SAP_000.pdf